CLINICAL TRIAL: NCT04441567
Title: Patient Reported Outcomes Measures Pilot Grant for Orthopedic Patients
Brief Title: Right-Size Clinic Visits Using Memora Platform for PROMIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: H-38859
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Orthopedic Disorders
Keywords: PROM; PROMIS; Memora Health Text messaging platform; SMS (Short Message Service); Orthopedic conditions; Recovery curves; Right-size clinic visits; CAT; SMS
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: This is a two-phase pilot study recruiting approximately 1500 subjects in each of the two phases. Phase 1 - No intervention, create recovery curves only. Phase 2 - Adjust clinic follow-up based on patient responses in relation to recovery curves generated from Phase 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (No Intervention): Participants in phase 1 will be observed and data about their recovery time will be collected from which recovery curves will be calculated for Phase 2
- Phase 2 (Experimental): Participants in Phase 2 will have their clinic visits potentially revised based on the phase 1 recovery curves which may increase or decrease the number of clinic visits they receive based on the PROMs reported.
  Interventions: Other: Right-size clinic visits

INTERVENTIONS:
Other: Right-size clinic visits — The curve created in Phase 1 will be used to guide the number of clinic visits based on PROMs reported by the participants in Phase 2.
  Arms: Phase 2

SUMMARY:
Developing novel methods of patient communication is crucial in providing value-based care to orthopedic patients. Healthcare technology platforms have been developed to improve patient communication methods particularly for the administration of patient-reported outcome measures (PROMs). However, the majority of these interventions rely on web-based platforms that require patients to have computer access. Among American households earning less than $30,000 per year, only 59% have access to a desktop or laptop and just 47% have broadband internet at home compared to mobile phone penetration which is estimated at 95% of which 93% regularly use text messages. The use of phone messaging may be the most effective means to have patients complete PROMs.

The Patient-Reported Outcomes Measurement Information System (PROMIS) is an NIH-funded, clinically validated method of tracking patient-reported outcomes to efficiently assess patient health status. PROMIS utilizes Item Response Theory (IRT) and computerized adaptive testing (CAT) to improve measurement precision and decrease survey time as compared to traditional PROMs.

The purpose of this two-phase study is to utilize Memora Health's text-messaging platform to collect web-based PROMIS CAT surveys from patients (Phase 1) and use this information to right-size clinic visits (Phase 2).

DETAILED DESCRIPTION:
Phase 1 will be a prospective evaluation of patients with the conditions listed. After consent, participants will complete PROMIS CAT questionnaires on their mobile phones to assess health status. During enrollment, participants will choose a method of completing the surveys throughout the duration of the study. The participants will either 1) receive a short message service(SMS) with a secure weblink to complete these PROMIS CAT questionnaires on a secure website, or 2) engage in two-way SMS communication by answering the survey questions individually by texting back their answers. The investigators will explain that the desired method of participation is by weblink due to privacy issues associated with two-way texting. The frequency at which the questionnaires will be sent is condition-specific. All patients will be seen in clinic at standard follow up time-points and will be asked to complete PROMIS questionnaires during each clinic visit, identical to the delivery of surveys while at home. The PROMIS measures collected over a 1-year period will be used to develop patient-based recovery curves.

Phase 2 will begin at the end of Phase 1 and compare each participant's recovery (based on the PROMs) against the established recovery curve that was generated in Phase 1 for their orthopedic condition. The investigators will right-size in-person clinic visits based on individual recovery as compared with expected recovery. Earlier clinic appointments will be given to participants at risk for a poor outcome (defined as any PROMIS score ≥1 standard deviation below the mean). All other participants will receive a phone call to make sure that participants feel they are doing well and to have any issues addressed. If it is felt that a visit is warranted, it will be recommended, and if a subject wishes to have a visit it will be scheduled. If the subject is happy with their progress, then that in-person clinic visit will be deferred until the next standard follow-up visit and the same process will occur. Some in-person visits will be mandatory when a physical exam or x-ray is required for optimal care. These are condition specific. For all participants, a final in-person follow-up visit will occur unless the subject is happy and does not want to be seen in person.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that are classified by the Current Procedural Terminology/International Classification of Diseases (CPT/ICD)-10 Diagnosis Codes, having sustained the injury within 3 weeks of enrollment for non-operative treatment or will undergo surgery during the enrollment period:
* Ankle Fracture
* Distal Radius Fracture
* Tibial Plateau Open reduction internal fixation (ORIF)
* Spine Operative

  * Anterior cervical discectomy with fusion (ACDF)
  * Cervical Laminectomy
  * Lumbar Fusion
  * Lumbar Decompression
* Spine Non-operative

  * Lumbar Stenosis
  * Lumbar Degenerative Disc Disease
* Rotator Cuff Repair
* Anterior cruciate ligament (ACL) Reconstruction
* Have personal use of cellular phone with access to the internet
* Speak either English or English as a primary language:

Exclusion Criteria:

* Limited and non-readers
* Vulnerable populations - incarcerated patients
* Patients with no cell phone to use for scoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Right-size clinic visits for specific orthopedic conditions | 2 years
  Right-size clinic visits for patients recovering at/better than expected while maintaining or improving overall patient-reported outcomes (PROMS) will be assessed by comparing to the mean condition-specific recovery curve from phase 1. Earlier clinic visits will be scheduled for those who are more than 1 standard deviation from the mean recovery at any time point and less frequent visits for all others to establish the right size clinic visits.
Patient-based recovery curves for specific orthopedic conditions | 1 year
  Each participant's recovery (based on the patient-reported outcome measures- PROMs) for their orthopedic condition will be assessed against the established recovery curve that was generated in phase one of the research for their condition.

SECONDARY OUTCOMES:
Average number of PROMs collected through SMS and weblink | 1 year
  The number of PROMs collected through SMS and weblink will be assessed. PROMs are standardized, validated questionnaires completed by patients to measure their perception of their functional well-being and health status.
Average number of PROMs collected during clinic visits | 1 year
  The number of PROMs collected during clinic visits will be assessed. PROMs are standardized, validated questionnaires completed by patients to measure their perception of their functional well-being and health status.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tornetta III, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No